CLINICAL TRIAL: NCT05408195
Title: Evaluate E-Care Acceptability for Older People Undergoing Chemotherapy at Home
Brief Title: E-Care Acceptability for Older People Undergoing Chemotherapy
Acronym: ONCO-CHATBOT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The use of CHATBOT is limited in the service for multiple reasons and nursing resources have been limited for several months, with no prospect of improvement in the months to come.
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/19/0517
Record Dates: First submitted 2022-05-24; First posted 2022-06-07 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: older adults; nurses; smartphones; chemotherapy; geriatric oncology.
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHATBOT users (Experimental): patients downloading and using the CHATBOT
  Interventions: Device: CHATBOT use

INTERVENTIONS:
Device: CHATBOT use — Patients benefiting from chemotherapy with outpatient follow-up (conventional follow-up by telephone calls) have the possibility to receive a weekly remote questionnaire (by email or SMS) via a CHATBOT on any terminal. This automated questionnaire collects data (completed by the patient and/or their caregivers) on tolerance and compliance to the care plan.

SUMMARY:
The main objective of this pilot study is to evaluate the acceptability of clinical data collection using a semi-automated e-solution based on the use of text messaging among older adults undergoing chemotherapy treatment at home.

DETAILED DESCRIPTION:
Most cancer diagnosis are made among the 70 years and over population. In this population, negative consequences of cancer treatments are of great concern, especially for those who are socially isolated or live in rural areas. International oncology societies recommend personalized treatments to reduce adverse events. However, few tools have been validated in this population to monitor compliance and risks of outpatient treatments. In addition, health professionals continue to manage unplanned patient calls which could disrupt effectiveness of their work. Our hypothesis is that the semi-automated collection of health data (text message questionnaires) during outpatient chemotherapy secures the patient's care pathway and optimizes care time, in particular for patients' education and support. Therefore, patients (and/or their caregivers) who benefit from calls follow-up (usual care), would have the possibility of receiving an additional weekly remote questionnaire (by email or SMS) via a CHATBOT on any terminal. This automated questionnaire collects data on tolerance and compliance with care plan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 70 years of age or older;
* Subjects undergoing chemotherapy treatment after a cancer diagnosis;
* Subjects managed by the oncogeriatrics team at the Toulouse University Hospital as part of an outpatient follow-up and followed by conventional telephone calls and CHATBOT support.

Exclusion Criteria:

* Patient's refusal to participate.
* Patient does not have sufficient equipment for downloading and using the CHATBOT tool
* Participant under guardianship, curatorship or safeguard of justice.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance of semi-automated follow-up | 6 months of CHATBOT use
  Proportion of patients who uploaded the application, Proportion of patients who received at least one questionnaire, Proportion of patients who answered at least one questionnaire, Completion questionnaire rate and answered questionnaire rate

CONTACTS AND LOCATIONS:
Overall Officials: Antoine PIAU, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No